CLINICAL TRIAL: NCT03806829
Title: Pilot Study: The Acute Effects of Commercially Available Drinks on the Endothelial Function of Humans Following a High-fat Meal
Brief Title: The Acute Effects of Commercially Available Drinks on the Endothelial Function of Humans Following a High-fat Meal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Highlands and Islands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ETHSHE1376
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Endothelial Dysfunction
Keywords: antioxidants; polyphenols; flow-mediated dilatation
MeSH Terms: interventions — Water; Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Water + Meal (Active Comparator): 250 ml Water and a high calorie, high fat meal (>900 kcal, 50g fat)
  Interventions: Other: Water
- Red Wine + Meal (Experimental): 250 ml Red Wine and a high calorie, high fat meal (>900 kcal, 50g fat)
  Interventions: Other: Red Wine
- Green Tea + Meal (Experimental): 250 ml Green Tea and a high calorie, high fat meal (>900 kcal, 50g fat)
  Interventions: Other: Green Tea
- Orange Juice + Meal (Experimental): 250 ml Orange Juice and a high calorie, high fat meal (>900 kcal, 50g fat)
  Interventions: Other: Orange Juice

INTERVENTIONS:
Other: Water — 250 ml
  Arms: Water + Meal
Other: Red Wine — 250 ml
  Arms: Red Wine + Meal
Other: Green Tea — 250 ml
  Arms: Green Tea + Meal
Other: Orange Juice — 250 ml
  Arms: Orange Juice + Meal

SUMMARY:
High fat diets are associated with impaired endothelial function and increased cardiovascular disease risk amongst our population. These negative effects are likely caused by triglyceride induced suppression of nitric oxide, which is produced from the endothelium, and/or an increase in oxidative stress.

Interestingly, previous studies have found that some beverages that are high in polyphenols and antioxidants may suppress the impairment in endothelial function observed following high fat meals/diets. Typically, these studies have investigated the ingestion of red wine, orange juice or green tea on outcome measures (typically flow mediated dilatation (FMD) of the brachial artery). Despite this previous research, no study has compared the effects of different beverages on endothelial outcomes following a high-fat meal within the same participants.

ELIGIBILITY:
Inclusion Criteria:

* Females to be postmenopausal and not on hormone replacement therapy
* 25 > BMI < 35
* Sedentary to light activity lifestyle.

Exclusion Criteria:

* History of cardiovascular disease (Hypertension, Atherosclerosis, endothelial issues etc).
* History of diabetes (Type 1 or type 2)
* Vegan or with food allergies or intolerances.
* Taking any antioxidants over the counter (Vit C, E or polyphenol supplements)
* Taking prescription medication for hypertension.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Endothelial (dys)function | 2 hours post-prandial
  Assessed via flow mediated dilatation

SECONDARY OUTCOMES:
Plasma Nitrite | 2 hours post-prandial
Plasma antioxidant capacity | 2 hours post-prandial
  Plasma oxygen radical absorbance capacity
Plasma ox-LDL | 2 hours post-prandial

CONTACTS AND LOCATIONS:
Overall Officials: Ian Megson, Megson, Principal Investigator — University of the Highlands and Islands
Locations (1):
- University of the Highlands and Islands, Inverness, United Kingdom

IPD SHARING:
Plan to Share IPD: No